CLINICAL TRIAL: NCT03813017
Title: Comprehensive Assessment of Subclinical Atherosclerosis in Patients With Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Osamah Hussein, Head of Internal Medicine A, Ziv Hospital
Other Study IDs: 0123-18-ZIV
Record Dates: First submitted 2019-01-13; First posted 2019-01-23 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Cardiovascular Diseases; Rheumatoid Arthritis; Atherosclerosis, Coronary
MeSH Terms: conditions — Cardiovascular Diseases; Arthritis, Rheumatoid; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular disease is a leading cause for morbidity and mortality in general population. The incidence of cardiovascular disease and their poor outcome is well documented in a broad spectrum of connective tissue diseases, especially in rheumatoid arthritis (RA). The risk of incident CVD is increased by 48% in patients with RA compared to the general population.

RA is associated with 50% increase in the mortality in patients with cardiovascular disease (CVD). One reason is the more frequent cardiovascular risk factors in RA patients compared with the general population. Patients with RA have a high risk of premature cardiovascular disease (CVD). The aim of the present study is to assess whether there are non-invasive measures that might predict arteriosclerosis in RA patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old (except for women till 75 years old)
2. Absence of established CVD:

   * Myocardial Infarction p/h
   * PCI with balloon and/or stent
   * Intermittent claudication
   * PAD / intervention
   * CAS /intervention
3. Signed informed consent form
4. Documented diagnosis of rheumatoid arthritis

Exclusion Criteria:

1. Known CVD
2. Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in Ziv Medical Center, Safed, Internal Medicine Department A, on 100 patients with rheumatoid artheritis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular disease risks in patient with theumatoid arthritis | 6 months
  Prediction of cardiovascular risks and proposed preventive treatment